CLINICAL TRIAL: NCT01801865
Title: Clinical Use of a New Neonatal MRI System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-2850
Record Dates: First submitted 2012-07-25; First posted 2013-03-01 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Magnetic Resonance Imaging
Keywords: NICU; MRI; Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI for Neonates (Experimental): All participants will receive an MRI in the NICU scanner in the GE OPTIMA 1.5T MRI at CCHMC.
  Interventions: Device: GE OPTIMA MR430s with HDX/GE Electronics

INTERVENTIONS:
Device: GE OPTIMA MR430s with HDX/GE Electronics
  Other Names: GE OPTIMA 1.5T MRI

SUMMARY:
The purpose of the present study is to make medically indicated state of the art/high end magnetic resonance imaging (MRI) exams available to all infants in the Cincinnati Children's Hospital Medical Center (CCHMC) Neonatal Intensive Care Unit (NICU).

DETAILED DESCRIPTION:
The current practice of transferring infants from the Neonatal Intensive Care Unit (NICU) to radiology departments and imaging in adult-sized magnetic resonance imaging (MRI) scanners is associated with significant safety and image quality issues. For these reasons, the smallest and/or sickest neonates are typically precluded from receiving an MRI exam. The overreaching goal of our research effort is to bring high-performance MRI into the NICU so that all neonates can benefit from the same quality of diagnostic imaging as adults. To accomplish this, we have converted a commercial small-bore 1.5 Tesla (T) MRI scanner designed for orthopedic use into a neonatal MRI system optimized for whole body imaging of neonates. To expand the imaging capabilities of the NICU MRI system, the measurement control electronics and operating system software of the FDA cleared imaging OPTIMA platform have been augmented with state of the art HDX electronics and software currently used on a conventional commercially available adult sized whole body MRI scanner. The clinical safety of the integrated HDX/OPTIMA NICU MRI system and its ability to produce diagnostic image quality has been shown in 15 pilot patients (CCHMC Protocol 2011-2045). The present protocol builds and expands upon the previous to use the integrated NICU MRI system to perform MRI exams in the neonatal population.

ELIGIBILITY:
Inclusion Criteria:

* Any infant admitted to the NICU at CCHMC
* Have a medical condition for which an MRI exam is indicated, as determined by the attending neonatologist
* Able to maintain body temperature for at least 90 minutes without the aid of an incubator or radiant warmer int he opinion of the attending neonatologist
* Parental/LAR permission obtained

Exclusion Criteria:

* Infants too large to fit in the customized NICU MRI system comfortably (expected to be infants heavier than 6 kg)
* Standard MRI exclusion criteria as set forth by the CCHMC Division of Radiology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2012-04; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth M Kline-Fath, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- NICU, Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The attending neonatologist determined whether the MRI scan was done with or without sedation. If possible, infants were scanned without sedation. Infants were prepared for the MRI exam by switching all monitoring devices over to MRI compatible monitors and provided with hearing protection.
Groups:
- MRI for Neonates: MRI
  GE OPTIMA MR430s with HDX/GE Electronics: MRI scan
Period: Overall Study
Arm/Group | MRI for Neonates
Started | 657
Completed | 615
Not Completed | 42
Not completed — Patients scanned on another MRI scanner | 35
Not completed — Physician Decision | 7

BASELINE CHARACTERISTICS:
Arm/Group | MRI for Neonates
Number analyzed (Participants) | 615
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 615
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: days] | 18.25 [0 to 156.95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280
  Male | 335
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Anatomy scanned [Count of Participants; unit: Participants]
  Abdomen | 7
  Orbit/Face/Neck | 7
  Pelvis and Extremity | 2
  Brain and Chest | 7
  Brain and Abdomen | 2
  Brain | 517
  Brain and Spine | 41
  Spine | 23
  Chest and Spine | 1
  Chest | 5
  Spine and Pelvis | 2
  Pelvis | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as Observed During and After Scanning.
Description: Any observed physical changes either related or not related to the MRI was recorded during and after scanning.
Time Frame: Day 1
Population: All patients have undergone clinically indicated and ordered MRI's.
Measure: Count of Participants; unit: Participants
Arm/Group | MRI for Neonates
Number analyzed (Participants) | 615
Participants | 4

2. Secondary Outcome: Each Infant's Baseline Measurement for Weight Will be Recorded to Ensure the Infant is Less Than 6 kg.
Description: These measures will be used in order to facilitate future design of coils and transport tables for the customized MRI system.
Time Frame: Day 1
Population: All patients have undergone clinically indicated and ordered MRI's.
Measure: Count of Participants; unit: Participants
Arm/Group | MRI for Neonates
Number analyzed (Participants) | 615
Participants | 615

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | MRI for Neonates
All-Cause Mortality (participants affected / at risk) | 0/615
Serious Adverse Events (participants affected / at risk) | 0/615
Other Adverse Events (participants affected / at risk) | 4/615
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI for Neonates (N=615)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Apneic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sedative therapy (Surgical and medical procedures) | 1 (1) — The patient received 2 doses of PO versed. The patient recovered, no sequelae. The event was related to clinically indicated sedation given to the subject for a clinically indicated scan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT01801865/Prot_000.pdf